CLINICAL TRIAL: NCT01631786
Title: Synchrotron Imaging of Human Ovaries Ex Situ
Status: Completed | Type: Observational
Sponsor: University of Saskatchewan (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Angela Baerwald, Assistant Professor, University of Saskatchewan
Other Study IDs: CIHR-THRUST-ARB-001
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Abnormal Female Reproductive Function
Keywords: Ovaries; Imaging; Ultrasonography; Synchrotron; Histology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — surgically removed human ovarian tissues and Formalin-fixed human ovarian tissues
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preserved ovaries: Ovaries or ovarian segments that have been fixed in 10% Formalin
- Fresh/non-preserved ovaries: Ovaries that have been surgically removed and placed in sterile saline

SUMMARY:
Ultrasonography is currently the most common diagnostic tool for imaging the female reproductive tissues. However, clinical ultrasonography is limited to the detection of ovarian structures ≥ 2 mm, with an inability to image microanatomy including small antral follicles and oocytes. The objective of this study is to determine whether the synchrotron can be used to effectively image bovine and human ovaries ex situ. We hypothesize that synchrotron imaging will provide greater resolution and thereby allow the detection of fine structural details of the ovary compared to conventional ultrasonography. Ovaries will be imaged using conventional ultrasonography, synchrotron and histology. We anticipate that our results will provide important information about ovarian physiology which can be applied to the study of female reproductive dysfunctions.

DETAILED DESCRIPTION:
The objective of our research is to determine whether the synchrotron is an effective tool for imaging human ovaries ex situ. Approximately 1 in every 6 women in Canada is affected by infertility; however, the underlying causes remain largely unknown. Imaging techniques are essential for increasing our understanding of normal and abnormal female reproductive biology. At present, ultrasonography is the most commonly-used tool to image human ovaries. However, ultrasonography only allows the detection of structures ≥ 2 mm in size within the ovaries, limiting the ability to detect smaller anatomic details (eg. the eggs and the surrounding cells and 'follicles' or the small fluid filled sacs that contain the eggs). Other limitations of ultrasonography for imaging the ovaries include a limited depth of penetration within the pelvis and the inability to see the ovaries clearly due to bowel activity and/or gas.

The synchrotron has been effectively used for imaging soft tissues, including the breast, heart and lungs. We hypothesize that the synchrotron will provide greater resolution for imaging the ovaries compared to conventional ultrasonography. Specifically, we anticipate that synchrotron imaging will provide greater structural details of the ovaries (including small follicles <2 mm and eggs) compared to conventional ultrasonography.

The study will consist of three different phases listed below:

* Phase 1 - Imaging of 10 fresh and preserved bovine ovaries
* Phase 2 - Imaging of 5 preserved human ovaries from the Department of Pathology
* Phase 3 - Imaging of 2-4 fresh human ovaries from women having their ovaries surgically removed

The initial imaging of bovine ovaries will help us determine the best synchrotron settings to image the human samples. All ovaries will be preserved using formaldehyde. In all 3 study phases, ovarian specimens will be imaged first with 2D and 3D ultrasonography and then with the Biomedical Imaging and Therapy Beamline (BMIT) at the Canadian Light Source. Furthermore, histologic sections of structures of interest within the ovaries will be made, and digital images will be acquired.

We believe that synchrotron imaging of human ovaries ex situ will be an important first step to develop future high-resolution tools for imaging reproductive tissues in situ.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing unilateral/bilateral oophorectomy at Saskatoon City Hospital or Royal University Hospital between May - August 2012

Exclusion Criteria:

* none

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in the Saskatoon Health Region
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Follicular counts | July-Aug 2012
  total number of antral ovarian follicles will be counted in the ultrasonographic and synchrotron images

SECONDARY OUTCOMES:
Diameter measurements | July-Aug 2012
  The diameters of ovarian follicles, cell layers of the follicle wall, corpora lutea, and cumulus oocyte complexes will be measured using ultrasonographic, synchrotron and histologic images
Microanatomy of ovarian tissues | July -Aug 2013
  Qualitative and quantitative evaluations of ovarian microanatomy using histology. Histological evaluations will be compared with synchrotron images.

CONTACTS AND LOCATIONS:
Overall Officials: Angela R Baerwald, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Canadian Light Source, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Singh J, Adams GP, Pierson RA. Promise of new imaging technologies for assessing ovarian function. Anim Reprod Sci. 2003 Oct 15;78(3-4):371-99. doi: 10.1016/s0378-4320(03)00100-3. PMID 12818654